CLINICAL TRIAL: NCT06089889
Title: Investigating the Impact of Ice Application on the Venous Puncture Pain in the Pediatric Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Sidra Sultan, Principal investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VPP RCT 001
Record Dates: First submitted 2023-10-03; First posted 2023-10-19 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Venous Puncture Pain
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Children will be allocated in two groups by randomization (lottery method). one group will be intervention group and other group would be control group
Who Masked: Outcomes Assessor
Masking Description: a staff nurse will be nominated for recording the child's pain intensity on video for objectively assessing the child's pain score.
  video recorder will be blinded of intervention. The staff nurse responsible for videotaping will be kept uninformed about the intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 will receive ice application as intervention 3 minutes before venous puncture.
  Interventions: Other: ice application
- Group 2 (Experimental): Group 2 will be control group, without ice application.
  Interventions: Other: control group

INTERVENTIONS:
Other: ice application — * Group 1 will undergo the first intervention, which involves the application of ice.
  * Ice pack will be applied on the site of venipuncture prior to intravenous procedures for 3 minutes.
  * The procedure of venous puncture will be carried out in accordance with established standard operating procedures (SOPs).
  * pain will be assessed through Wong baker Faces Pain scale immediate after venous puncture procedure.
  after taking consent from parents/guardians, the pain response of children will be video taped for the purpose of objectively assessing the pain. and data will be kept confidential.
  Arms: Group 1
Other: control group — * Group 2 will be control group, which involves no ice application
  * The venipuncture procedure will be carried out according to established standard operating procedures (SOPs), pain will be assessed by Wong Baker Faces Pain Scale immediate after venous puncture procedure.
  After obtaining consent from parents/guardians, the pain responses of children will be videotaped for the purpose of objectively assessing pain, and the data will be kept confidential.
  Arms: Group 2

SUMMARY:
the goal of this RCT is: "To evaluate the effectiveness of a non-pharmacological method (ice application) in reducing venous puncture pain among children aged 5 to 7 years.".

An (RCT) will be conducted, involving 114 children, a non-probability convenience sampling will be used and children will randomly assign to two groups by lottery method. One group will receive ice application as an intervention, while other group will be control group, having no ice application.

DETAILED DESCRIPTION:
Children often undergo venous punctures in wards and emergency rooms, a procedure that is both painful and distressing for both children and their parents. When pain is not effectively managed, it can lead to fear, anxiety, uncooperative behavior, unsuccessful attempts, prolonged procedure duration, and overall dissatisfaction with the care provided. Various methods, both pharmacological and non-pharmacological, can help reduce pain during venous puncture, but most of these preparations are not feasible in urgent situations due to their time-consuming nature. The aim of this study is to evaluate the effectiveness of a non-pharmacological method (ice application) in reducing venous puncture pain in children. It is hypothesized that there is a significant difference in the pain intensity/score among children in the intervention group (ice application) and the control group (without ice application).

The rationale of this study is to find a cost-effective method for reducing pain during IV puncture, minimizing hospitalization costs for children, and alleviating their fear of pain. A randomized controlled trial (RCT) will be conducted, involving 114 children. Non-probability convenience sampling will be used, and children will be randomly assigned to two groups using the lottery method. One group will receive ice application as an intervention, while the other group will serve as the control group. The effectiveness of this approach will be assessed through a comparative analysis of these two groups. The study will span a duration of 3 months, starting after the synopsis receives approval. The target population for the study will be children aged 5 to 7 years. Pain will be assessed using the Wong-Baker Faces Pain Rating Scale. Data will be analyzed using SPSS version 24. Descriptive statistics (frequency, percentage) will be used to describe the characteristics of the study population. The Chi-square test will be used to examine the demographic information of the two groups. Independent t-tests will be used to compare the means of both groups after intervention. The significance level of the tests will be considered at a p-value < 0.05. The anticipated findings of this study lie in its comprehensive analysis of this methodology to determine the most economically feasible non-pharmacological approach. By focusing on resource-limited hospitals in Pakistan, the study aims to swiftly identify a method that can be readily implemented, effectively cutting down hospitalization costs for children while also addressing their pain-related issues. This research not only establishes a crucial benchmark in evidence collection but also paves the way for addressing pain-related challenges linked to venipuncture in pediatric patients, offering substantial benefits in the long run

ELIGIBILITY:
Inclusion Criteria:

* Children within age group of 5-7 years
* Children who were advised to undergo venous puncture in the pediatric ward

Exclusion Criteria:

* Chronically ill
* Mentally handicapped
* Already having local anesthesia at the venous puncture site

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
venous puncture pain | pain will be assessed immediate after venous puncture procedure, and data collection will take 2 months
  pain will be measured by Wong baker faces pain scale after venipuncture.Donnie Wong and Connie Baker developed The Wong-Baker Faces Pain Rating Scale in 1983. They research that children had difficulty rating their pain with numbers yet responded well to facial expressions. Consequently, they developed the scale to help children better communicate their pain. The Wong-Baker Faces Pain Rating Scale is a tool that aids individuals in expressing their physical pain. It employs facial expressions, numerical values, and descriptive words, allowing for varied ways to convey pain intensity. This self-assessment method encompasses a range of six faces, from a smiling face denoting "no hurt" (0) to a tearful face representing "hurts worst" (10), enabling effective communication of pain severity.
  The Wong-Baker Faces Pain Scale has been extensively studied in literature, with its reliability and validity having already been established for children aged 3 to 18 years

IPD SHARING:
Plan to Share IPD: No